CLINICAL TRIAL: NCT07087522
Title: Impact of Preprocedural Stress Ball Use on Radial Artery Outcomes in Elective Coronary Angiography: A Randomized Controlled Trial
Brief Title: Impact of Preprocedural Stress Ball Use on Radial Artery Outcomes in Elective Coronary Angiography
Acronym: SPARROW
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Emre Eynel, MD, Dr. Emre Eynel, Specialist in Cardiology, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SEAH-2025-SPARROW-001
Record Dates: First submitted 2025-06-16; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Coronary Arterial Disease (CAD); Radial Artery Spasm; Radial Artery Occlusion; Transradial Angiogram; Visual Analog Pain Scale
Keywords: Radial Artery; Radial Artery Spasm; Radial Artery Occlusion; Coronary Anjiography; Transradial Approach; Hand Exercise; Stress Ball; Vascular Complications
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the intervention group (stress ball use) or the control group (standard care) in a parallel design, with no crossover between groups.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Both the interventional cardiologist performing the radial procedure and the outcome assessor conducting the Doppler ultrasonography will be blinded to the participant's group allocation. This double-blind design aims to minimize procedural and assessment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress Ball Group (Experimental): Participants will perform hand exercises using a stress ball for 5 minutes, 3 times per day, for 3 consecutive days prior to radial angiography.
  Interventions: Behavioral: Stress Ball Use
- Control Group (No Intervention): No hand exercise or stress ball use will be applied before radial angiography.

INTERVENTIONS:
Behavioral: Stress Ball Use — Participants will perform hand exercises using a rubber stress ball for 5 minutes, 3 times daily, for 3 days prior to radial angiography.
  Arms: Stress Ball Group

SUMMARY:
This randomized, double-blind, controlled trial aims to evaluate the effect of preprocedural hand exercise using a stress ball on the incidence of radial artery spasm and other vascular complications in patients undergoing elective coronary angiography via the transradial approach. A total of 400 adult patients scheduled for elective diagnostic or interventional coronary procedures will be randomly assigned to either an intervention group (preprocedural stress ball exercise) or a control group (standard care). The intervention group will perform hand exercises with a soft stress ball for 5 minutes, three times daily, for three consecutive days prior to the procedure.

The primary outcomes are the incidence of radial artery spasm during the procedure and the overall rate of radial artery complications.

Secondary outcomes include patient-reported pain score (visual analog scale) during the procedure and the incidence of radial artery occlusion at 7 days, assessed by Doppler ultrasonography.

This study aims to determine whether this simple, low-cost strategy can reduce radial artery-related complications and improve patient comfort during transradial coronary procedures.

DETAILED DESCRIPTION:
Radial artery access has become the preferred approach for coronary angiography and percutaneous coronary intervention (PCI) due to its superior safety profile, reduced bleeding complications, earlier patient mobilization, and improved overall comfort compared to the traditional femoral approach. Despite these advantages, transradial procedures are not entirely free of complications. Radial artery spasm (RAS) remains a significant concern, with reported incidence rates ranging from 4% to 20%, depending on operator experience and patient-related factors. Additionally, vascular complications such as hematoma, arterial dissection, pseudoaneurysm, bleeding at the access site, and post-procedural radial artery occlusion (RAO) can affect procedural success and may limit future access via the same route.

Handgrip exercise has been proposed as a simple, non-invasive, and cost-effective strategy to improve arterial compliance, increase vessel diameter, and potentially reduce vasospasm by enhancing endothelial function and promoting local vasodilation. Despite promising physiologic rationale and preliminary findings in other settings (such as arterial diameter augmentation prior to AV fistula creation), the role of preprocedural hand exercise in preventing radial artery complications during coronary procedures has not been systematically studied in a randomized controlled trial.

This single-center, randomized, double-blind, controlled clinical trial aims to assess whether regular preprocedural hand exercise using a soft stress ball can reduce the incidence of RAS and vascular complications in patients undergoing elective coronary angiography via the transradial approach.

A total of 400 adult patients (aged 18 to 85 years), scheduled for elective diagnostic or interventional coronary procedures via the radial artery, will be enrolled. Patients with contraindications to radial access, prior significant upper limb vascular disease, or inability to perform the hand exercise regimen will be excluded.

Participants will be randomly assigned in a 1:1 ratio to either the intervention group or the control group using a computer-generated randomization sequence. Both the interventional cardiologist performing the procedure and the clinical staff responsible for outcome assessment will remain blinded to group allocation.

Intervention Group: Patients will be instructed to perform handgrip exercises using a soft stress ball for 5 minutes per session, three times per day, for three consecutive days prior to the procedure. Adherence will be monitored through a patient-completed exercise log and direct interview at the time of hospital admission.

Control Group: Patients will receive standard preprocedural care without any specific hand exercise recommendations.

The primary outcomes of the study include:

Incidence of radial artery spasm, defined clinically by resistance to catheter advancement, patient-reported discomfort, or the need for pharmacologic spasmolytics during the procedure.

Overall rate of vascular complications, including access site hematoma, arterial dissection, pseudoaneurysm, and access-related bleeding.

The secondary outcomes include:

Patient-reported pain during radial access, measured using the Visual Analog Scale (VAS).

Incidence of radial artery occlusion (RAO), evaluated at 7 days post-procedure via Doppler ultrasonography.

This study seeks to determine whether a brief period of structured, low-intensity hand exercise can serve as an effective adjunct to routine preprocedural care in patients undergoing transradial coronary angiography. If proven effective, this strategy could be incorporated into standard practice, offering a low-risk and widely applicable method to enhance procedural outcomes, minimize patient discomfort, and preserve radial artery integrity for future access.

Additionally, this trial will contribute valuable data to the growing field of procedural preparation optimization, focusing on patient-involved, non-pharmacological interventions that promote vascular health and procedural success.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years
* Elective radial coronary angiography planned
* Written informed consent provided
* Ability to understand and comply with the stress ball exercise protocol (3×5 minutes/day for 3 days prior to procedure)
* Palpable radial pulse on the planned access site

Exclusion Criteria:

* Emergent or urgent coronary procedures
* Known radial artery occlusion or non-palpable radial pulse on the intended access side
* Prior arteriovenous fistula or vascular surgery in the ipsilateral arm
* History of Raynaud's disease, severe peripheral artery disease, or Buerger's disease
* Neurological or musculoskeletal disorders affecting hand grip (e.g., stroke, advanced arthritis, peripheral neuropathy)
* Cognitive impairment or psychiatric condition preventing protocol adherence
* Inability to use hand muscles effectively (e.g., recent hand trauma, paralysis)
* Unwillingness or inability to perform the stress ball exercises as instructed
* Pregnancy or breastfeeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Radial Artery Spasm Rate | Periprocedural
  Incidence of periprocedural radial artery spasm as reported by the operator, characterized by catheter resistance, patient discomfort, or vasodilator need.
Pain Score During Procedure (VAS) | Immediately after the procedure
  Visual Analog Scale (VAS) score reported by the patient (0 = no pain, 10 = worst pain imaginable).

SECONDARY OUTCOMES:
Radial Artery Occlusion (RAO) | 7 days after the procedure
  Radial artery occlusion confirmed by color Doppler ultrasonography. RAO is defined as the absence of flow in the radial artery at the puncture site, assessed in both longitudinal and transverse views.
Radial Artery Cannulation Duration | During radial artery cannulation procedure
  Total time from radial sheath insertion, measured in minutes.
Number of Puncture Attempts | During radial artery cannulation procedure
  Number of needle punctures required for successful access.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University Training and Research Hospital, Sakarya, Adapazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The de-identified individual participant data (IPD) will be made available upon reasonable request after publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication of the primary results.
Access Criteria: Qualified researchers with a methodologically sound proposal and appropriate institutional ethics approval may request access to the data. A formal data-sharing agreement must be signed. Requests will be reviewed and approved by the principal investigator (Dr. Emre Eynel).

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-18): https://cdn.clinicaltrials.gov/large-docs/22/NCT07087522/Prot_SAP_000.pdf